CLINICAL TRIAL: NCT03539562
Title: Therapeutic Rest to Delay Admission in Early Labor: A Prospective Study on Morphine Sleep
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 17-21855
Record Dates: First submitted 2018-02-27; First posted 2018-05-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Labor Pain; Early Labor
MeSH Terms: conditions — Labor Pain; Obstetric Labor, Premature | interventions — Morphine; Promethazine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Accepted Morphine Sulfate: Patients accepted morphine and promethazine as a method for pain management in early or prodromal labor.
  Interventions: Drug: Morphine Sulfate and Promethazine
- Declined Morphine Sulfate: Patients declined morphine and promethazine as a method for pain management in early or prodromal labor.

INTERVENTIONS:
Drug: Morphine Sulfate and Promethazine — Morphine sulfate and promethazine
  Other Names: Morphine Sleep
  Groups: Accepted Morphine Sulfate

SUMMARY:
This will be a prospective study on labor characteristics, and obstetric and neonatal outcomes in women who accept and women who decline morphine as a form of pain management in labor. The study will also investigate patient satisfaction with this form of analgesia. The participants will be those who accept morphine and promethazine and those who decline morphine and promethazine for pain control.

DETAILED DESCRIPTION:
Objective: Therapeutic rest in labor involves administration of parenteral analgesics in early or prodromal labor to relieve the patient's discomfort and allow for progression of labor while the patient rests. No prospective studies exist which examine the safety and clinical utility of therapeutic rest in early labor, and no published studies examine the potential benefits of therapeutic rest from the perspective of either patient satisfaction or cost-effectiveness. The investigators aim to determine whether therapeutic rest using morphine and promethazine is associated with variations in labor characteristics, or obstetric or neonatal outcomes as well as patient satisfaction with this form of pain management.

Methods: This will be a prospective cohort study. Women who are eligible for therapeutic rest (reactive non-stress test, normal amniotic fluid, in prodromal or early labor as defined by obstetric provider, and plan to discharge home after evaluation) will be recruited for the study. Participants will receive routine obstetric care by providers who are unaware of patient enrollment. A research assistant will then approach all participants in the postpartum period, prior to discharge from the hospital or with a phone call if permitted by the patient, to complete a questionnaire including patient satisfaction items. Chart review will be performed to determine differences in hospital stay and common obstetric and neonatal outcomes to compare these data among women who do and do not choose to receive therapeutic rest. These results will provide insight into a common clinical practice, helping to not only guide management at institutions where therapeutic rest is commonly utilized but also potentially encourage its initiation at hospitals were therapeutic rest is not available.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies between 37w0d and 41w6d gestation
* Presentation to triage for rule out labor as primary indication and found to be in early labor
* Offered therapeutic rest by obstetric provider with plan to discharge home after evaluation

Exclusion Criteria:

* Allergy to morphine sulfate or promethazine
* Being without an attendant to safely transport the patient home
* Present to triage for other indication (decreased fetal-movement, premature rupture of membranes, hypertension, etc.)
* Multiple gestation
* Known fetal anomaly
* Placenta previa, active maternal Herpes Simplex Virus disease, or any other contraindication to vaginal delivery
* Recommendation for direct admission to L&D for maternal or fetal indication.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women presenting to Labor & Delivery Triage who meet inclusion criteria and are offered morphine sulfate and promethazine by labor provider for therapeutic rest.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
The proportion of women who were admitted in active labor (6 cm or greater cervical dilation). | 0 hours to 2 weeks
  Admission in active labor

SECONDARY OUTCOMES:
Time in hours between the start of contractions to being offered therapeutic rest | 1-2 weeks after delivery
  Duration of contractions in hours before presenting for rule out labor
Time in hours between being offered therapeutic rest and admission to labor and delivery | 1-2 weeks after delivery
  Latency period between being offered therapeutic rest and admission
Time in hours between admission to labor and delivery and complete cervical dilation | 1-2 weeks after delivery
  Length of admission
Time in hours between admission to labor and delivery and birth time | 1-2 weeks after delivery
  Length of admission
Time in hours between complete cervical dilation and birth time | 1-2 weeks after delivery
  Length of second stage
Proportion of women who required induction of labor | 1-2 weeks after delivery
  Induction of labor
Proportion of women who required augmentation of labor | 1-2 weeks after delivery
  Augmentation of labor
Proportion of women who received an epidural | 1-2 weeks after delivery
  Epidural use
Type of delivery | 1-2 weeks after delivery
  Mode of delivery
Proportion of women diagnosed with chorioamnionitis | 1-2 weeks after delivery
  Presence of maternal infection
APGAR scores of neonate | 1-2 weeks after birth
  Neonatal clinical assessment
Umbilical cord gas values | 1-2 weeks after birth
  Neonatal laboratory assessment
Proportion of newborns admitted to Intensive Care Nursery | 1-2 weeks after birth
  Neonatal Intensive Care Unit admission
Neonatal Intensive Care Unit length of stay in days | 1-2 weeks after birth
  Length of stay in the Intensive Care Nursery
Proportion of women with meconium present during labor | 1-2 weeks after delivery
  Presence of meconium
Patient responses (yes or no) to a 4-question survey conducted after delivery to determine satisfaction with morphine and promethazine as a form of therapeutic rest. | 1-4 weeks after delivery
  Patient satisfaction assessment

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Gaw, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center at Mission Bay, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] ACOG Committee Opinion #295: pain relief during labor. Obstet Gynecol. 2004 Jul;104(1):213. PMID 15229040
- [Background] Mackeen AD, Fehnel E, Berghella V, Klein T. Morphine sleep in pregnancy. Am J Perinatol. 2014 Jan;31(1):85-90. doi: 10.1055/s-0033-1334448. Epub 2013 Mar 7. PMID 23471604
- [Background] Koontz WL, Bishop EH. Management of the latent phase of labor. Clin Obstet Gynecol. 1982 Mar;25(1):111-4. doi: 10.1097/00003081-198203000-00015. PMID 7067192
- [Background] S G. Obstetrics: Normal and Problem Pregnancies. 5th ed. Philadelphia, PA: Churchill Livingstone; 2007.
- [Derived] Maykin MM, Ukoha EP, Tilp V, Gaw SL, Lewkowitz AK. Impact of therapeutic rest in early labor on perinatal outcomes: a prospective study. Am J Obstet Gynecol MFM. 2021 May;3(3):100325. doi: 10.1016/j.ajogmf.2021.100325. Epub 2021 Feb 2. PMID 33545440